CLINICAL TRIAL: NCT04998422
Title: Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of HG381 as Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study of HG381 Administered to Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HitGen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HG381CN101
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: HG381 Monotherapy Dose Escalation Cohort (Experimental): Subjects will receive HG381 IV at every one week intervals (Q1W). Escalating doses of HG381 will be evaluated by the traditional 3+3 design.
  Interventions: Drug: HG381
- Part B: HG381 Monotherapy Dose Expansion Cohort (Experimental): Subjects will be administered the recommended Phase 2 dose of HG381 IV Q1W established in Part A of the study.
  Interventions: Drug: HG381

INTERVENTIONS:
Drug: HG381 — HG381 is available as white to off-white cake or powder for solution for injection at a unit dose strength of 5 mg per vial. HG381 will be administered as IV injection.
  Other Names: HG381 for Injection

SUMMARY:
This is a Phase I, first in human, open-label, non-randomized, multicenter study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, preliminary efficacy and establish a recommended dose of HG381 administered intravenously (IV) alone in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
The trial consists of a dose escalation phase and a cohort expansion phase.In dose escalation phase, escalating doses of HG381 will be evaluated as guided by the traditional 3+3 design . In cohort expansion phase, subjects will receive HG381 alone at a single dose level determined based on the data form dose escalation phase. In total, approximately 57 subjects will participate in the study, approximately 42 in the dose-escalation cohort, and approximately 15 in the expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Life expectancy of at least 3 months.
* Histological or cytological documentation of an advanced solid tumor，subjects with advanced/recurrent solid tumors, who have progressed on, be intolerant of, or ineligible for, all available therapies for which clinical benefit has been established.
* Measurable disease per RECIST version 1.1, there is at least one measurable lesion during the screening period.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Adequate organ function : Hematologic system: Hemoglobin ≥9 g/dL, Absolute neutrophil count [ANC] ≥1.5x10^9/L, Platelets ≥100x10^9/L, INR ≤ 1.5 and APTT ≤1.5 x ULN; Hepatic system: Total bilirubin ≤1.5 x ULN, ALT and AST ≤ 2.5 x ULN; Renal system: serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (calculated by the Cockcroft-Gault formula); Cardiac system: left ventricular ejection fraction (LVEF) ≥50% ; QT interval (QTcF) ≤470 ms for women, and ≤450 ms for men; Endocrine system: Thyroid-stimulating hormone (TSH) is within the normal limits.
* Subjects with fertility must agree to take medically approved effective contraceptive measures during the entire trial period and at least 3 months after the last medication.

Exclusion Criteria:

* Chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anticancer therapy within 4 weeks.
* Concurrent medical condition requiring the use of other systemic immunosuppressive treatment within 4 weeks before the first dose of study treatment.
* Receipt of any live vaccine within 4 weeks of the start of study treatment.
* Receipt of unmarketed clinical trial drugs or treatments within 4 weeks of the start of study treatment.
* Receipt of surgery or interventional treatment (excluding tumor biopsy, puncture, etc.) within 4 weeks of the start of study treatment.
* History or evidence of cardiovascular and cerebrovascular diseases risk.
* Subjects with uncontrolled diabetes.
* Symptomatic central nervous system (CNS) metastases or asymptomatic CNS metastases that have required steroids within 2 weeks prior to first dose of study treatment.
* Currently or in the past suffering from malignant tumors.
* Uncontrollable pleural effusion, pericardial effusion or ascites still need to be drained frequently after appropriate intervention.
* Active or suspected autoimmune disease.
* History of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia, or evidence of active, non-infectious pneumonitis.
* Toxicity from previous treatment including: Toxicity Grade ≥3 related to prior immunotherapy and that led to study treatment discontinuation; Toxicity related to prior treatment that has not resolved to Grade ≤ 1.
* Subjects who have acute bacterial, viral or fungal infections and require systemic anti-infective treatment.
* Positive test for syphilis antibodies or human immunodeficiency virus (HIV) antibodies.
* Subjects who are allergic to test drugs and excipients.
* Women who are pregnant or breastfeeding.
* Known drug or alcohol abuse.
* Patients with mental or neurological diseases.
* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Subjects who have a history of serious systemic disease or any other reason are not suitable to participate in this trial as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | Up to Day 21
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
Maximum Tolerated Dose (MTD) | Up to 12 months
  The maximum tolerated dose (MTD) is defined as the maximum dose where the number of cases of DLT ≤ 1/6 of the total number of cases during the DLT observation period. At least 6 evaluable subjects are required to determine MTD.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
  An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or requires medical judgement.
Severity of AEs | Up to 24 months
  The severity of AEs will be graded utilizing the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of HG381 | Up to 12 months
  Up to 42 patients with advanced/metastatic solid tumors will be enrolled in Dose Escalation to determine the RP2D of HG381 as monotherapy.
Best objective response based on RECIST 1.1 | Up to 24 months
  Best objective response rate is defined as the percentage of subjects with a best overall confirmed CR or PR at any time as per disease-specific criteria.
HG381 concentrations in plasma following administration of HG381 alone | Cycle 1 Days 1, Cycle 2 Days 1 and Cycle 3 Days 1: pre-infusion and at multiple time points (up to 24 hours) post-infusion (Cycle length=21 days)
  Blood samples will be collected at indicated time points for plasma pharmacokinetic (PK) analysis of HG381.
Maximum observed concentration (Cmax) following administration of HG381 alone | Cycle 1 Days 1, Cycle 2 Days 1 and Cycle 3 Days 1: pre-infusion and at multiple time points (up to 24 hours) post-infusion (Cycle length=21 days)
  Blood samples will be collected at indicated time points for plasma PK analysis following administration of HG381 monotherapy.
Area under the concentration-time curve (AUC) following administration of HG381 alone | Cycle 1 Days 1, Cycle 2 Days 1 and Cycle 3 Days 1: pre-infusion and at multiple time points (up to 24 hours) post-infusion (Cycle length=21 days)
  Blood samples will be collected at indicated time points for plasma PK analysis following administration of HG381 monotherapy.
Apparent terminal phase half-life (t½) following administration of HG381 alone | Cycle 1 Days 1, Cycle 2 Days 1 and Cycle 3 Days 1: pre-infusion and at multiple time points (up to 24 hours) post-infusion (Cycle length=21 days)
  Blood samples will be collected at indicated time points for plasma PK analysis following administration of HG381 monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, M.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- HitGen Inc., Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Zhu Y, An X, Zhang X, Qiao Y, Zheng T, Li X. STING: a master regulator in the cancer-immunity cycle. Mol Cancer. 2019 Nov 4;18(1):152. doi: 10.1186/s12943-019-1087-y. PMID 31679519
- [Background] Liu S, Cai X, Wu J, Cong Q, Chen X, Li T, Du F, Ren J, Wu YT, Grishin NV, Chen ZJ. Phosphorylation of innate immune adaptor proteins MAVS, STING, and TRIF induces IRF3 activation. Science. 2015 Mar 13;347(6227):aaa2630. doi: 10.1126/science.aaa2630. Epub 2015 Jan 29. PMID 25636800
- [Background] Barber GN. STING: infection, inflammation and cancer. Nat Rev Immunol. 2015 Dec;15(12):760-70. doi: 10.1038/nri3921. PMID 26603901
- [Background] Abe T, Barber GN. Cytosolic-DNA-mediated, STING-dependent proinflammatory gene induction necessitates canonical NF-kappaB activation through TBK1. J Virol. 2014 May;88(10):5328-41. doi: 10.1128/JVI.00037-14. Epub 2014 Mar 5. PMID 24600004
- [Background] Ramanjulu JM, Pesiridis GS, Yang J, Concha N, Singhaus R, Zhang SY, Tran JL, Moore P, Lehmann S, Eberl HC, Muelbaier M, Schneck JL, Clemens J, Adam M, Mehlmann J, Romano J, Morales A, Kang J, Leister L, Graybill TL, Charnley AK, Ye G, Nevins N, Behnia K, Wolf AI, Kasparcova V, Nurse K, Wang L, Puhl AC, Li Y, Klein M, Hopson CB, Guss J, Bantscheff M, Bergamini G, Reilly MA, Lian Y, Duffy KJ, Adams J, Foley KP, Gough PJ, Marquis RW, Smothers J, Hoos A, Bertin J. Design of amidobenzimidazole STING receptor agonists with systemic activity. Nature. 2018 Dec;564(7736):439-443. doi: 10.1038/s41586-018-0705-y. Epub 2018 Nov 7. Erratum In: Nature. 2019 Jun;570(7761):E53. doi: 10.1038/s41586-019-1265-5. PMID 30405246
- [Background] Sivick KE, Desbien AL, Glickman LH, Reiner GL, Corrales L, Surh NH, Hudson TE, Vu UT, Francica BJ, Banda T, Katibah GE, Kanne DB, Leong JJ, Metchette K, Bruml JR, Ndubaku CO, McKenna JM, Feng Y, Zheng L, Bender SL, Cho CY, Leong ML, van Elsas A, Dubensky TW Jr, McWhirter SM. Magnitude of Therapeutic STING Activation Determines CD8+ T Cell-Mediated Anti-tumor Immunity. Cell Rep. 2019 Oct 15;29(3):785-789. doi: 10.1016/j.celrep.2019.09.089. No abstract available. PMID 31618645
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774